CLINICAL TRIAL: NCT00053612
Title: Prevention of HIV Shedding in Women - Trial of Vitamin A
Brief Title: Vitamin A to Reduce HIV in Vaginal Secretions and Prevent Viral Transmission
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01AI343844; R01-AI343844
Record Dates: First submitted 2003-02-03; First posted 2003-02-05 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2007-08

CONDITIONS: HIV Infections; Vitamin A Deficiency; HIV Seronegativity
Keywords: HIV-1; Women; Vitamin A; Shedding
MeSH Terms: conditions — HIV Infections; Vitamin A Deficiency | interventions — Vitamin A

INTERVENTIONS:
Drug: Vitamin A

SUMMARY:
HIV infected individuals with vitamin A deficiency may be more likely to transmit the virus to others than HIV infected individuals who have normal levels of vitamin A. The presence of HIV DNA in vaginal secretions may indicate a greater risk for transmission of HIV to others. The purpose of this study is to determine if taking vitamin A decreases the level of HIV DNA in vaginal secretions.

DETAILED DESCRIPTION:
Vitamin A deficiency leads to pathological changes in mucosal epithelium, including the vagina, and is correlated with immune dysfunction in both HIV-1 infected and uninfected individuals. Recent studies of genital tract shedding of HIV-1 DNA in infected women have found that lower serum concentrations of vitamin A were strongly associated with detection of HIV-1 in vaginal secretions. In addition, maternal vitamin A deficiency has been associated with significantly increased risk of vertical HIV-1 transmission. This study will assess the effect of vitamin A supplementation on the prevalence and quantity of HIV-1 DNA and RNA in cervical and vaginal secretions.

Participants in this study will be HIV infected nonpregnant women in Mombasa, Kenya. Participants will be randomized to receive 6 weeks of daily dosage of either 10,000 IU vitamin A or placebo. Cervical and vaginal swabs will be obtained at enrollment and at Week 6 for detection and quantification of HIV-1 DNA and RNA. In addition, venous blood will be obtained at the two time points for quantification of plasma HIV-1 RNA, CD4 lymphocyte count, and serum vitamin A levels.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected

Exlusion Criteria:

* Pregnant

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan Kreiss, MD, MPH, Principal Investigator — Universiy of Washington, Seattle, WA